CLINICAL TRIAL: NCT06624943
Title: Evaluating the Impact of Introducing Basaglar, a Long-acting Analog Insulin, on Clinical and Quality of Life Outcomes in Youth with Diabetes in Mali
Brief Title: Introducing Biosimilar Insulin Glargine to the Treatment Regimen of Children and Youth with Type 1 Diabetes in Mali
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Life for a Child Program, Diabetes Australia (Other)
Collaborators: Sante Diabete Mali (Other); Hospital of Mali (Unknown); Centre Hospitalier du Luxembourg (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/27/CE/USTTB; #2208-05490 (Other Grant/Funding Number: The Leona M. and Harry B. Helmsley Charitable Trust)
Record Dates: First submitted 2024-09-29; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: children; adolescents; insulin glargine; Mali
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (No Intervention): Continue current treatment with either intermediate- and short-acting human insulin, or pre-mixed insulin, both via needle and syringe
- Intervention (Experimental): Switched to once daily injection of biosimilar insulin glargine via reusable pen and three mealtime bolus insulin injections of short-acting human insulin via needle and syringe
  Interventions: Drug: biosimilar insulin glargine

INTERVENTIONS:
Drug: biosimilar insulin glargine — Once daily injection of biosimilar insulin glargine via reusable pen
  Other Names: Basaglar
  Arms: Intervention

SUMMARY:
This study aimed to evaluate the impact on blood glucose control and quality of life in children and youth with type 1 diabetes in Mali by switching the insulin regimen from human insulin via needle and syringe, to long-acting biosimilar insulin glargine delivered by reusable pens combined with short-acting insulin via needle and syringe.

DETAILED DESCRIPTION:
Analog insulins are widely used in middle- and high-income countries. However, use of analog insulin remains limited in lower-income countries due to their increased cost and lack of access, and human insulin remains the mainstay of treatment in these settings.

Long-acting (basal) analog insulin such as glargine have the benefit of a longer duration (up to 24 hours) and a minimal peak action, and generally, only one injection per day is required. Although glargine insulin has been shown to reduce the risk of overnight hypoglycemia, consistent improvement in blood glucose control (measured by HbA1c) when compared to human insulin has not been shown, and its impact on quality of life is also inconclusive. Furthermore, these studies have all been done in highly resourced countries.

Life for a Child (LFAC) has been providing diabetes supplies (insulin, syringes, meters and strips for blood glucose self-monitoring), diabetes-related education, mentoring and technical support to Santé Diabète in Mali since 2008. In 2021, LFAC commenced supplying Basaglar (glargine) insulin with insulin pen devices (HumaPen Ergo ll). This provided a unique opportunity to investigate the effect of introducing glargine (Basaglar) insulin in the low-resource setting of Mali, one of the world's poorest countries.

ELIGIBILITY:
Inclusion Criteria:

(i) diagnosed with T1D in accordance with World Health Organization criteria

(ii) duration of T1D ≥12 months at time of enrolment

(iii) aged <25 years at time of enrolment

(iv) current insulin regimen consisting of Humulin NPH® and R, or pre-mixed insulin (30/70 R/NPH), with no prior use of analogue insulin

(vi) willing to regularly self-monitor blood glucose (SMBG) levels ≥2 times a day with a blood glucose meter and strips

(vii) live in or within one hour's travelling distance of Bamako

Exclusion Criteria:

(i) Previous use of analog insulin

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 260 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
HbA1c | Baseline, 3-, 6-, 9- and 12-month follow-up visits
  HbA1c was measured at each study time point using point of care testing via a Siemens DCA calibrated to international standards (DCA Vantage™ Analyzer (Siemens Healthcare Diagnostics, Tarrytown NY, US)). For HbA1c readings >14% (>130 mmol/mol), the maximum reading of this analyser, HbA1c was recorded as 14% (130 mmol/mol).

SECONDARY OUTCOMES:
Episodes of diabetic ketoacidosis | Baseline, 3-, 6-, 9- and 12-month follow-up visits
  Diabetic ketoacidosis was defined as hyperglycaemia (BGL>11mmol/L/200mg/dL) with a venous pH<7·3 or serum bicarbonate <15mmol/L and ketonuria and/or ketonaemia
Episodes of severe hypoglycaemia | Baseline, 3-, 6-, 9- and 12-month follow-up visits
  Severe hypoglcaemia was defined as an event with severe cognitive impairment (with or without coma and convulsions) requiring assistance by another person to administer carbohydrates, glucagon, or intravenous dextrose to restore glycaemia
Diabetes Quality of Life in Youth - Short Form | Baseline, 6- and 12-month follow-up visits
  The 21-item Diabetes Quality of Life in Youth - Short Form scale (TC Skinner et al., Diabetologia 2006; 49, 621-628) was administered to participants in both study arms To assess the psychosocial impact of their respective insulin treatment regimens
Participant self-reported satisfaction (intervention arm only) | 12-month follow-up visit
  A 5-item structured questionnaire was administered to participants in the intervention group to evaluate their satisfaction with the new insulin regimen, experience of using reusable insulin pens, and their experience of hypo- and hyperglycaemic episodes over the study period
Feedback from local HCPs on implementation of the study intervention | At 12 months
  A 6-item questionnaire was administered to HCPs at the end of the study, to obtain feedback on the training they received, their confidence in teaching youth and families on switching to the new insulin regimen, and opinion on its impact on hypo- and hyperglycaemic episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Besançon, MSC, Principal Investigator — ONG Santé Diabète,Bamako,Mali & Unité PACRI,Conservatoire National des Arts et Métiers,Paris,France
Locations (1):
- Hôpital du Mali, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No
Due local privacy regulations, individual de-identified participant data will not be shared.